CLINICAL TRIAL: NCT02383719
Title: Oro-nasal Mask Patient Comfort Evaluation
Brief Title: A Feasibility Study Evaluating the Use of a Non-invasive Ventilation Mask
Acronym: mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Convergent Engineering, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Conveng - 002
Record Dates: First submitted 2015-02-27; First posted 2015-03-09 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Noninvasive Ventilation; Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

ARMS (1):
- Oro-nasal mask (Experimental): All patients are included in this arm. Patients in this group receive the experimental oro-nasal mask during non-invasive ventilation
  Interventions: Device: Oro-nasal Mask

INTERVENTIONS:
Device: Oro-nasal Mask

SUMMARY:
Evaluate the clinicians assessment of the use of an oro-nasal mask during non-invasive ventilation (non-intubated) with a feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* patient requiring non-invasive ventilation in an intensive care unit

Exclusion Criteria:

* patient not stable for non-invasive ventilation
* patient with unprotected airway
* excessive secretions
* patient with facial surgery
* agitated patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Alnuaimat, M.D., Principal Investigator — University of Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Comfort of mask fit for patients receiving non-invasive ventilation at Shands hospital in Gainesville Florida
Groups:
- Oro-nasal Mask: Oro-nasal Mask
Period: Overall Study
Arm/Group | Oro-nasal Mask
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oro-nasal Mask
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Clinician Assessment of Use With a Questionnaire
Description: With the questionnaire we desired to discern the clinicians perception of use of the experimental oro-nasal mask. The questionnaire featured the ease of installation, the ease of use, and the perceived comfort of the patient. Each of the scores were on a scale from 1-5 and each were recorded to be used for individual assessment. Thus each patient has multiple assessment scores individually reported as outcomes.
  The clinicians were asked on a scale of 1-5 please rate their agreement with the statements The mask was easy to use. 1 strongly disagree, 2 somewhat disagree, 3 neutral, 4 somewhat agree, 5 strongly agree Your perception of patient comfort was acceptable. 1 strongly disagree, 2 somewhat disagree, 3 neutral, 4 somewhat agree, 5 strongly agree
Time Frame: During non-invasive ventilation with the oro-nasal mask
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Oro-nasal Mask: All patients in this group received the experimental oro-nasal mask for evaluation of use. Patient's received non-invasive ventilation were switched to this mask upone study initiation.
Arm/Group | Oro-nasal Mask
Number analyzed (Participants) | 18
units on a scale
  Ease of Use | 5 [4 to 5]
  Patient Comfort | 4 [4 to 5]

ADVERSE EVENTS:
Arm/Group | Oro-nasal Mask
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No